CLINICAL TRIAL: NCT00001867
Title: Effect of Pregnancy on Uveitis
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990179; 99-EI-0179
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-09

CONDITIONS: Postpartum Period; Pregnancy; Uveitis
Keywords: Cytokine; Gestation; Postpartum; Pregnancy; Th 1 Lymphocyte; Th 2 Lymphocyte; Uveitis
MeSH Terms: conditions — Uveitis

SUMMARY:
The purpose of this study is to gain information about the course of uveitis (a type of eye inflammation) during pregnancy and the postpartum period (six months after delivery). Some reports have indicated the condition may improve or disappear without treatment during pregnancy and recur postpartum, requiring treatment. No systematic studies have been done, however, to examine a link between pregnancy and disease suppression.

All medicines for uveitis have side effects-particularly for pregnant women, their unborn babies, and breast-feeding mothers. The information gained may help guide treatment decisions for these patients in the future.

Women who are between 2 and 20 weeks pregnant and have had uveitis within 2 years of becoming pregnant will be followed monthly with an eye examination and blood tests until six months after giving birth. The eye examination will include dilation of the pupils to look at the back of the eye. Photos of the eye will be taken to record changes that occur due to uveitis. The blood tests will assess immune function and try to determine whether levels of hormones and cytokines are related to uveitis disease activity. Patients who develop an inflammation and significant vision loss may require treatment, possibly with eye drops or injections near the eye. Treatment will be decided in consultation with the patient's obstetrician.

DETAILED DESCRIPTION:
Pregnancy is thought to be associated with the remediation of some disease and exacerbation of other conditions. Anecdotal case reports suggest that uveitis may remit or improve during pregnancy and recur in the postpartum period. This observation is supported by findings in an experimental autoimmune uveitis model in mice. We propose to study the natural history of ocular inflammation in a series of pregnant women who have had ocular inflammation (uveitis) in the two year period prior to becoming pregnant. Women will be enrolled between 2 and 20 completed weeks of gestation at which time they will receive a complete ophthalmologic examination and will have blood drawn for cytokine and hormone evaluation. These procedures will be repeated at monthly intervals until 6 months postpartum. Treatment of uveitis will ensue as medically indicated and in consultation with the woman's obstetric care provider. The goal of this investigation is to determine whether cytokine levels are correlated with disease expression. Such information may be useful to inform decisions about how to best manage pregnant and postpartum uveitis patients in the future.

ELIGIBILITY:
Females with a history of unilateral or bilateral immune-mediated, non-infectious inflammatory ocular disease that required topical and/or systemic immunosuppresive medications at least once in the past two years or who are currently under treatment for unilateral or bilateral non-infectious ocular inflammation and having diagnosed uveitis, scleritis, or autoimmune corneal disorders in the past two years.

First and second trimester pregnancy.

Informed consent from the patient.

No pregnancy complications which require medical treatment and special obstetric care.

No hematolgical disorder that would preclude blood draws for investigational purposes.

No current ocular or systemic infection.

No current malignancy.

No current endocrine disorders.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 1999-09; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wegmann TG, Lin H, Guilbert L, Mosmann TR. Bidirectional cytokine interactions in the maternal-fetal relationship: is successful pregnancy a TH2 phenomenon? Immunol Today. 1993 Jul;14(7):353-6. doi: 10.1016/0167-5699(93)90235-D. PMID 8363725
- [Background] Raghupathy R. Th1-type immunity is incompatible with successful pregnancy. Immunol Today. 1997 Oct;18(10):478-82. doi: 10.1016/s0167-5699(97)01127-4. PMID 9357139
- [Background] Raghupathy R. Maternal anti-placental cell-mediated reactivity and spontaneous abortions. Am J Reprod Immunol. 1997 Jun;37(6):478-84. doi: 10.1111/j.1600-0897.1997.tb00263.x. PMID 9228305